CLINICAL TRIAL: NCT05786196
Title: Multicenter Glaucoma Study Investigating Standalone Canaloplasty, Randomized Controlled Trial: iTrack Advance (Nova Eye, Inc.) Compared to OMNI (Sight Sciences)
Brief Title: Multicenter Glaucoma Study Investigating Standalone Canaloplasty
Acronym: MAGIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Eye, Inc. (Industry)
Collaborators: Nova Eye Medical GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NE 05021
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Primary Open Angle Glaucoma
Keywords: Canaloplasty
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- iTrack Advance (Active Comparator): Ab-interno canaloplasty utilizing the iTrack Advance microcatheter device (Nova Eye, Inc.)
  Interventions: Device: Ab-interno canaloplasty utilizing the iTrack Advance device
- OMNI Surgical System (Active Comparator): Ab-interno canaloplasty utilizing the OMNI Surgical System
  Interventions: Device: Ab-interno canaloplasty utilizing the OMNI Surgical System

INTERVENTIONS:
Device: Ab-interno canaloplasty utilizing the iTrack Advance device — 360 degree microcatheterization and viscodilation of Schlemm's canal
  Arms: iTrack Advance
Device: Ab-interno canaloplasty utilizing the OMNI Surgical System — 360 degree microcatheterization and viscodilation of Schlemm's canal
  Arms: OMNI Surgical System

SUMMARY:
A multicenter, randomized, clinical trial to evaluate the efficacy of canaloplasty performed as a standalone procedure using the iTrack™ Advance canaloplasty device (Nova Eye, Inc.) as compared to the OMNI® Surgical System (Sight Sciences) in patients with mild to moderate primary open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 22 years or older at the time of surgery
* Diagnosed with mild to moderate primary open angle glaucoma
* Candidate for canaloplasty surgery: i.e., catheterization of Schlemm's canal and subsequent viscodilation of Schlemm's canal, without trabeculotomy
* Intolerance to medical therapy OR need/willingness to reduce medications
* At the Screening Visit, IOP of ≤ 30 mmHg while on 1-4 ocular hypotensive medications
* At the Baseline Visit, unmedicated IOP ≥ 21mmHg and ≤ 36 mmHg, and ≥ 3mmHg higher than medicated IOP
* Shaffer grade of ≥ 3 in all four quadrants
* Central corneal thickness ≥ 480µm and ≤ 620 µm
* Able and willing to comply with the study procedures and attend all follow-up visits
* Understands and signs the informed consent

Exclusion Criteria:

* Any of the following prior treatments for glaucoma (study eye):

  1. Laser trabeculoplasty

     i. Selective Laser Trabeculoplasty (SLT) conducted within 6-months of the Screening Visit ii. Prior Argon Laser Trabeculoplasty
  2. iStent or iStent Inject within 180 days of the Screening Visit
  3. Endocyclophotocoagulation (ECP) or Micropulse laser
  4. Trabeculectomy or other bleb forming procedure including Xen, Express, and glaucoma draining device/valve
  5. Prior canaloplasty (ab interno and ab externo)
  6. Prior goniotomy, or trabeculotomy (ab externo and ab interno)
  7. Hydrus microstent
  8. Suprachoroidal stent (e.g., Cypass, iStent Supra, MINIject)
  9. Concurrent IOP-lowering procedure other than use of the iTrack Advance canaloplasty device OR the OMNI Surgical System at the time of surgery (e.g., ECP, CPC, etc.)
* Acute angle closure, traumatic, congenital, malignant, uveitic or neovascular glaucoma, pigmentary glaucoma or pseudoexfoliative glaucoma
* Cataract surgery within 6 months of the Screening Visit in the study eye
* History of fellow eye with cataract surgery within 30 days of Screening
* Subjects at significant risk by a washout of ocular hypotensive medication, and/or subjects where the unmedicated IOP is expected to exceed the upper limit of 36 mmHg
* Use of systemic medications (either current, within 30 calendar days of Screening exam, or anticipated) that may cause an increase in IOP, (e.g., systemic steroids including inhaled and oral steroids used on a regular basis)
* Ocular and/or systemic diseases that could affect the corneal endothelium (such as corneal endothelial dystrophy, intraocular inflammation and infection, or congenital abnormalities)
* History of penetrating keratoplasty or another corneal transplant
* BCVA of 20/200 or worse in the fellow eye not due to cataract
* Previous treatment with OMNI or iTrack (Note: permitted if fellow eye only was treated)
* BCVA of 20/50 or worse in the study eye not due to posterior capsular opacification

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The mean change in unmedicated Intraocular pressure (IOP) at Month-12 compared to baseline | 12 months
  IOP will be measured at each visit with Goldmann applanation tonometry
Percentage of eyes achieving a 20% or greater reduction in unmedicated Intraocular pressure (IOP) at Month-12 compared to baseline and without any other intervention (medication or secondary surgery) | 12 months
  IOP will be measured at each visit with Goldmann applanation tonometry

CONTACTS AND LOCATIONS:
Overall Officials: Shamil Patel, MD, MBA, Principal Investigator — Eye Physicians and Surgeons of Arizona
Locations (5):
- Breyer Kaymak Klabe Augenchirurgie, Düsseldorf, Germany
- Hospital Clinico San Carlos, Servicio de Oftalmologia, Madrid, Spain
- United Kingdom (3):
  - Princess Alexandra Eye Pavilion, NHS Lothian, Edinburgh
  - St. Paul's Eye Unit, Liverpool University, Liverpool
  - Manchester Royal Eye Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No